CLINICAL TRIAL: NCT01138215
Title: The Immunogenicity of Varicella-zoster Virus Vaccine in HIV-infected Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HIV-NAT 111
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Varicella-zoster Virus
Keywords: varicella-zoster virus vaccine; varicella-zoster virus antibody; immunogenicity; safety and efficacy; HIV-infected children; Assess protective VZV Antibody; Adverse events from VZV vaccine
MeSH Terms: conditions — HIV Infections; Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Receive 1 course of VZV vaccine : 2 doses of vaccines with 3 months apart.
  Interventions: Biological: VZV vaccination

INTERVENTIONS:
Biological: VZV vaccination — Dose : 0.5 ml Route : subcutaneous injection (SC)

SUMMARY:
To study about the immunogenicity, safety and efficacy of varicella-zoster virus vaccine in HIV-infected children.

DETAILED DESCRIPTION:
VZV causes two clinical diseases, primary infection results in varicella (chickenpox) after which virus latent in dorsal root ganglion. Reactivation of VZV results in herpes zoster (shingles) about years or decades. Immunocompetent children, varicella generally mild self limiting illness. In HIV infected children, VZV is often more severe illness with progressive varicella characterized by continuing eruption of lesions and high fever persist into second weeks, as well as encephalitis, hepatitis and pneumonia can developed. Zoster in immunocompromised patient become disseminated with lesions appearing outsides primary dermatomes and with visceral complications and can cause recurrences of herpes zoster. VZV illness in patients with immunodeficiency disorders require admission to hospital and the use of antiviral drugs. Sometimes, antiviral drug fails in immunocompromised children. Passive immunization with varicella zoster-immunoglobulin (VZIG), administered within three days of exposure, is effective in preventing disease or in reducing severity of illness in susceptible immunocompromised persons. About half of the cases of varicella in immunocompromised children occur without a recognised exposure to VZV. Both severe and fatal varicella has been documented despite appropriate immunoprophylaxis withVZIG. Furthermore, VZIG is expensive and short supply. These limitations make passive immunization a less than optimum strategy for preventing chickenpox. Permanent protection provided by administering the vaccine to high-risk persons would be preferable.

Sartori AM., University of Sao Paolo in Sep 2004 found that after give two doses of the varicella vaccine in 41 susceptible HIV-infected childrens in CDC class N1 or A1. Seroconversion occurred in 53% and 60% of vaccines after one and two doses, respectively. No significant fall in CD4 T lymphocytes or increase in HIV viral load at eight weeks after vaccination.

Saro H. Armenian, University of Southern California in Nov 2005 administrated single dose of live varicella vaccine to 10 HIV infected children. After vaccination, positive VZV-LPA response was detected in 50% of patients at week 2 and 100% at week 4, remained positive in 90% at week 52. VZV IgG was detected in 11% at week 2, 67% at week 8, only 33% at week 52.

Myron J. Levin, University of Colorado in June 2006-2008 study about the safety and immunogenicity of vaccine in varicella-zoster virus (VZV) naive, HIV-infected children with moderate symptoms and/or more pronounced past or current decreases in CD4+ T cell counts. Recipients (97 children) were stratified into 3 groups : group I - CDC category 1 and immunologic category 1 (least affected group of HIV-infected children), group II - CDC category A, B, or N and immunologic category 2 (CD4% = 15-24), group III : CDC category C and/or immunologic category 3, but at least 3 months prior to vaccination, had achieved clinical category A or N and equivalent of immunologic category 1 (CD4% = 25). After 2 doses of vaccines , 79% of children developed VZV-specific antibody and/or CMI 2 months after vaccine and 83% were responders 1 year after vaccination. Bekker V., Emma Children's Hospital, Netherland in Nov 2006 administered 2 doses of varicella vaccine to 15 VZV-seronegative HIV-1 infected children (total lymphocyte counts > 700 lymphocytes/microl) and 6 HIV-negative VZV-seronegative. Only 60% of the HIV-1 infected children had VZV-specific Ab after two immunizations, where as 100% of the siblings seroconverted.

Thai HIV infected children usually start antiretroviral late due to limited access to care with more severe suppressed of immune status than children in developed countries. Moreover, VZV vaccine is not in the country guideline and still expensive. We would like to provide VZV prevention for this group of children and to evaluate the VZV antibody response in Thai HIV children after VZV vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected children.
2. Aged between 1 to 15 years.
3. CD4 T lymphocyte percentage ≥ 15% or ≥ 200 cell/ml within 6 months at time of enrollment.
4. Written informed consent was obtained from each child's parent or guardian before enrollment.
5. HIV-infected children who age more than 7 years old sign assent.

Exclusion Criteria:

1. History of clinical varicella or zoster.
2. History of exposure to VZV within 1 month before study entry.
3. Received varicella vaccine.
4. Received immunoglobulin or blood product within 3 months before study entry.
5. Using oral steroid or immunosuppressive drugs within 3 months before study entry.
6. History of hypersensitivity to vaccine component (Neomycin).

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Proportion of children with protective VZV Antibody in HIV infected children after 2 doses of VZV vaccine. | 1 month after vaccine completion

SECONDARY OUTCOMES:
Adverse events from VZV vaccine. | 1 month after completion of vaccine
Compare proportion of children who developed VZV antibody by baseline characteristics e.g. immune status, age, gender. | 1 month after completion of vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org